CLINICAL TRIAL: NCT07040748
Title: Multimodal Immersive Virtual Reality Training for Improving Cognition in Adults With Metabolic Syndrome: A Randomized Clinical Trial
Brief Title: Immersive Virtual Reality Training for Improving Cognition in Adults With Metabolic Syndrome
Acronym: VIRTUAL-METS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Maite Garolera, Principal Investigator of the Brain, Cognition, and Behavior Research Group (C3-CST)., Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202316-10Fundació la MaratóTV3
Record Dates: First submitted 2025-05-28; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Cognitive impairment; Virtual Reality; Cognitive Training
MeSH Terms: conditions — Metabolic Syndrome; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two parallel groups: one receiving a multimodal group-based intervention using immersive virtual reality (Virtual-METS), and a control group receiving treatment as usual. The intervention consists of 24 sessions over 12 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Immersive VR-Based Multimodal Intervention (Virtual-METS) (Experimental): Participants in this arm will receive a multimodal group-based intervention using immersive virtual reality (IVR) without headsets. The intervention includes mindfulness (10 minutes), cognitive training (30 minutes), and physical exercises (20 minutes) delivered through MK360 immersive technology. Sessions are conducted in groups of 5 participants, twice per week for 12 weeks (24 sessions in total), led by a neuropsychologist.
  Interventions: Behavioral: Immersive VR-Based Multimodal Intervention (Virtual-METS)
- No Intervention: Treatment as Usual (Control Group) (No Intervention): Participants in this arm will continue with their usual care, including routine medical visits and remotely administered psychoeducational guidelines to support diet, physical activity, and adherence to pharmacological treatment. They will not receive any specific intervention during the study period.

INTERVENTIONS:
Behavioral: Immersive VR-Based Multimodal Intervention (Virtual-METS) — This intervention consists of a 12-week, group-based program using immersive virtual reality technology (MK360) without head-mounted displays. Each 60-minute session combines mindfulness practices adapted from the Mindfulness-Based Stress Reduction (MBSR) program, cognitive training targeting attention, processing speed, memory, and executive function through realistic virtual environments (such as parks, markets, or home interiors), and chair-based physical exercises focused on balance, stretching, and muscle strengthening. The intervention is delivered in small groups of five participants, twice per week, for a total of 24 sessions, and is led by a trained neuropsychologist.
  Arms: Experimental: Immersive VR-Based Multimodal Intervention (Virtual-METS)

SUMMARY:
This study aims to evaluate the effectiveness of a multimodal intervention using immersive virtual reality (Virtual-METS) to improve cognitive function in middle-aged adults with metabolic syndrome and subjective cognitive complaints. The intervention combines cognitive training and physical exercise in group sessions over 12 weeks.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS) has been associated with an increased risk of cognitive decline and potentially Alzheimer's disease. Given the high prevalence of MetS in older adult populations, there is an urgent need for alternative, non-pharmacological solutions to improve cognitive impairment associated with MetS. Immersive Virtual Reality (IVR) technology offers a unique opportunity to improve traditional interventions and accessibility for populations with physical, cognitive, or emotional constraints. The Virtual-METS project aims to evaluate the effects of a multimodal IVR intervention that combines cognitive training and physical exercise on eighty- four adults with MetS, aged between 45 and 70 years, and with subjective cognitive complaints. Participants will be randomly assigned to either the experimental group (Virtual-METS) or the control group (treatment as usual, TAU) in a single-blind, randomized clinical trial. The Virtual-METS intervention will be delivered in a group session with 5 participants, twice per week for 12 weeks (24 sessions). Measures of cognition, assessed by a neuropsychological battery and eye-tracking tasks (primary measures), as well as treatment compliance, functionality, and quality of life (secondary measures), will be assessed at baseline, post-treatment, and after 6 months. In addition, ophthalmologic examinations, carotid Doppler ultrasound, and a panel of blood-based and gut-derived biomarkers will be collected to explore physiological mechanisms underlying cognitive and clinical changes. An economic evaluation of cost-effectiveness, treatment costs, and quality-adjusted life-years, compared to TAU, will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrated criteria for the MetS: central obesity (waist circumference ≥ 94 cm for men or ≥ 80 cm for women) and at least 2 of the criteria described as follow: Triglycerides ≥ 150 mg/dl or specific treatment of this lipid disorder; HDL-C < 40 mg/dl (men) or < 50 mg/dl (women) or specific treatment of this lipid disorder; Systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85 mmHg or previously diagnosed hypertension treatment; Basal glycemia ≥ 100 mg/dl or type 2 diabetes previously diagnosed).
* Age: between 45 and 70 years old.
* Subjective cognitive complaints: Subjective Cognitive Decline Questionnaire (≥ 7).
* Ability to fully understand and speak Spanish or Catalan.

Exclusion Criteria:

* Confirmed or suspicion of dementia (MMSE<24).
* Diagnosis of severe psychiatric, neurological, developmental disorders, systemic pathologies, hematological, hormonal, nutritional pathology, and/or neoplasm that are known to cause cognitive deficits.
* Other severe comorbidities considered a probable bias for the study: a cardiac history of unstable angina, recent myocardial infarction within the last 3 months, congestive heart failure, significant heart valve dysfunction, or unstable hypertension; taking medications that could negatively affect cognitive function.
* Physical, motor, or sensory alterations that impede the neuropsychological examination or the rehabilitation program.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Differences between groups in scores of global cognition | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Global cognition is assessed with the Montreal Cognitive Assessment (MoCA) a screening tool designed to identify mild cognitive impairment (MCI) and other cognitive deficits. The MoCA takes around 10-15 minutes to complete and consists of 30 items (range=0-30). Higher scores mean a better outcome.
Differences between groups in scores of sustained attention | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Sustained attention is measured with the Test of Word Accentuation. Scores range from 0-30, higher scores mean a better performance.
Differences between groups in verbal memory | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Verbal memory is measured with the Auditory Verbal Learning Test (AVLT). It is a word-learning test where five presentations of a 15-word list are given, each followed by an attempted recall. This is followed by a second 15-word interference list (list B), followed by recall of list A. Delayed recall and recognition are also tested. For each trial, the score ranges from 0 to 15, with higher scores indicating better memory performance. The total learning score (sum of the five List A trials) ranges from 0 to 75. Delayed recall and recognition scores also range from 0 to 15. Higher scores indicate better verbal memory performance.
Differences between groups in scores of auditory attention | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Auditory attention is measured with Digit Span Forward (WAIS-IV). Participants are asked to repeat numbers in the same order as read aloud by the examiner. Scores range from 2 to 8, with higher scores indicating better attention span.
Differences between groups in scores of working memory | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Working memory is assessed using Digit Span Backward (WAIS-IV), where participants repeat number sequences in reverse order. Scores range from 2 to 8, with higher scores indicating better working memory.
Differences between groups in scores of processing speed | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Processing speed is measured with the Digit Symbol Coding subtest from the WAIS-III. It consists of replacing symbols that lack verbal meaning with numbers based on a key. Scores range from 0 to 133, with higher scores indicating better processing speed.
Differences between groups in scores of sustained attention and impulsivity | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Conners Continuous Performance Test - 3rd Edition (CPT-3) is task-oriented computerised assessment of attention-related problems. Participants are presented with a repetitive array of visual stimuli on a computer screen for 14 min. Participants are instructed to press the space bar every time a letter other than "X" appears and to not press the space bar when "X" appears. The rate of stimulus presentation varies according to 1, 2, and 4 s intervals throughout the task. Measures: Correct Detection (Higher rates indicate better outcome), Reaction times (Lower scores indicate better outcome), Omission errors (Lower rates indicate better outcome), and Commission errors (Lower rates indicate better outcome).
Differences between groups in scores of visuospatial memory | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Visuospatial memory is assessed with the Brief Visuospatial Memory Test - Revised (BVMT-R). Immediate memory is evaluated through the total score of three learning trials, with scores ranging from 0 to 36. Delayed memory is assessed through free recall (score range: 0 to 12) and recognition (number of correctly identified figures, corrected for false positives). Higher scores indicate better visuospatial memory performance.
Differences between groups in scores of logical memory | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Verbal episodic memory is assessed with Logical Memory I and II (WMS-IV), evaluating immediate and delayed recall of short stories. Scores range from 0 to 25 for each story, with a maximum total score of 50 when two stories are administered. In addition, a recognition phase is included, with scores ranging from 0 to 30. Higher scores across all components indicate better verbal episodic memory.
Differences between groups in scores of visual scanning and processing speed | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Visual scanning and processing speed are measured with the Trail-Making Test-A version. Participants are asked to connect a series of numbered circles on a page in numerical order. Completion time is recorded in seconds, with lower scores indicating better performance.
Differences between groups in scores of executive function and cognitive flexibility | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Executive functioning and cognitive flexibility are measured with the Trail-Making Test-B version. Participants are asked to connect a series of circles that contain both numbers and letters in alternating numerical and alphabetical order. Completion time is recorded in seconds, with lower scores indicating better performance.
Differences between groups in scores of executive functioning | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Executive functioning is assessed with the Modified Wisconsin Card Sorting Test (M-WCST), which evaluates abstract reasoning, cognitive flexibility, and the ability to shift problem-solving strategies. Performance is scored based on the number of categories completed, total errors, and perseverative errors. Higher scores in perseverative errors (range: 0 to >23) and total errors (range: 0 to >31) indicate worse performance, while more categories completed reflect better executive functioning (range: 0 to 8).
Differences between groups in scores of selective attention, inhibition, and processing speed | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Selective attention, inhibition, and processing speed are measured with the Stroop Color and Word Test. Participants are asked to name the color of a series of color patches (Stroop Color Naming), read a series of color words (Stroop Word Reading), and name the color of a series of color words where the word and color do not match (e.g., the word "red" written in blue ink), Stroop Color-Word Interference. Higher scores mean a better outcome.
Differences between groups in scores of phonetic fluency | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Phonemic verbal fluency is assessed using the PMR test, in which participants are asked to produce as many words as possible beginning with the letters P, M, and R, one minute per letter. The total score is the sum of all correct, non-repeated words across the three trials. Higher scores indicate better phonemic fluency and executive function.
Differences between groups in scores of semantic verbal fluency | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Semantic verbal fluency is assessed with a category fluency task in which participants are asked to name as many words as possible belonging to a specific semantic category (e.g., animals, fruits) within one minute. The total score is the number of correct, non-repeated words produced. Higher scores indicate better semantic fluency and lexical access.

SECONDARY OUTCOMES:
Differences between groups in Body Weight | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Body weight measured in kilograms, used as an indicator of metabolic status.
Differences between groups in waist circumference | Baseline, post-intervention (12 weeks), and 6-month follow-up
  Waist circumference measured in centimeters at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest. Indicator of abdominal fat.
Differences between groups in blood pressure | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Systolic and diastolic blood pressure measured in mmHg using an automated sphygmomanometer after 5 minutes of rest.
Differences between groups in fasting glucose | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Fasting glucose levels obtained from a venous blood sample after 8-12 hours of fasting. Indicator of glycemic control.
Differences between groups in lipid profile | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Lipid profile including total cholesterol, HDL, LDL, and triglycerides measured via fasting blood samples (milligrams per deciliter (mg/dL)).
Differences between groups in fasting insulin | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Serum insulin measured after overnight fasting using standardized immunoassay methods. Reflects insulin resistance.
Differences between groups in scores of functionality | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Functionality is measured with a 12-item World Health Organization Disability Assessment Schedule-II (WHODAS-II). Patients are asked to state the level of difficulty experienced, considering how they usually do the activity. The scale scores each item as "none" (1) to "cannot do" (5). The total score is calculated with an SPSS syntax, and the range varies from 0 to 100, with higher scores reflecting more significant disability.
Differences between groups in scores of quality of life | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Quality of Life is measured with EuroQol a self-completion questionnaire, which consists of five questions: covering mobility, hygiene, activities, pain, and anxiety. The descriptive system divides each of the 5 dimensions into three levels of response: the absence of a problem, some problem, and extreme problem. Lower scores indicate better outcomes. In addition, the questionnaire has a plus scale where the participants rated their health state on a scale of 0-100. In this scale, higher scores indicate better outcome.
  The WHOQOL-BREF assesses quality of life (QOL) within the context of an individual's culture, value systems, personal goals, standards and concerns.
Differences between groups in cognitive reserve | Baseline only.
  Cognitive reserve is assessed with the Cognitive Reserve Questionnaire, which evaluates factors such as education, occupation, and engagement in cognitive and social activities. Scores range from 0 to 24, with higher scores indicating greater cognitive reserve.
Expectation for treatment at baseline | Baseline only.
  Treatment expectations are assessed with the Expectation for Treatment Scale (ETS), a validated questionnaire that measures participants' beliefs and expectations about the potential benefits of the intervention. Total scores range from 5 to 25, with higher scores indicating more positive treatment expectations.
Differences between groups in subjective cognitive complaints | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Subjective cognitive complaints are measured using the MiCog questionnaire, which evaluates participants' perceived difficulties in daily cognitive functioning. Total scores range from 0 to 24, with higher scores indicating more cognitive complaints.
Differences between groups in general health status | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  General health is assessed using the Goldberg Health Questionnaire, a screening tool for psychological distress and general well-being. Higher scores indicating higher psychological distress.
Differences between groups in scores of depressive symptoms | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Depression is measured with the Patient Health Questionnaire-9 (PHQ-9) which scores each of the 9 DSM-IV criteria as "not at all" (0 points) to "nearly every day" (3 points). Total scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
Differences between groups in scores of anxiety symptoms | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Anxiety is measured with the 7-item Generalized Anxiety Disorder Scale (GAD-7), a Likert-type scale with questions ranging from "not at all" (0 points) to "nearly every day" (3 points). The maximum score is 24. Higher scores mean a worse outcome.
Differences between groups in healthy lifestyle habits | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Healthy lifestyle habits are evaluated using the Healthy Lifestyle Questionnaire, a validated Spanish-language instrument that evaluates physical activity, nutrition, and psychological well-being. Total scores range from 0 to 120, with higher scores indicating healthier lifestyle behaviors.
Differences between groups in sedentary behavior | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Sedentary behavior is measured with the short version of the Sedentary Behavior Questionnaire (SBQ-s), which asks about time spent in sedentary activities on weekdays and weekends. Total scores are reported in average hours per day, with higher values indicating greater sedentary behavior.
Differences between groups in scores of Sleep Quality | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Sleep Quality is measured with The Pittsburgh Sleep Quality Index (PSQI). This test presents 24 items, although only 19 are taken into account for the correction. This test is divided into 7 dimensions, namely, sleep quality, sleep onset latency, sleep duration, sleep efficiency, sleep disturbances, hypnotic drugs, and daytime dysfunction. Total scores range from 0 to 21, with higher scores indicating worse sleep quality.
Differences between groups in physical performance | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Physical performance is assessed using the Short Physical Performance Battery (SPPB), which includes balance, walking speed, and chair stand tests. Each component is scored from 0 to 4, and the total score ranges from 0 to 12, with higher scores indicating better physical function.
Differences between groups in carotid artery ultrasound measures | Baseline and 6-month follow-up.
  Intima-media thickness of the carotid arteries is measured using Doppler ultrasound to assess subclinical atherosclerosis.
Differences between groups in scores of eye-tracking data | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Eye-tracking tasks will measure cognitive processing through saccades, fixations, and pupil response during attention and memory tasks.
Differences between groups in intraocular pressure | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Intraocular pressure (IOP) measured in both eyes using Goldmann applanation tonometry (millimeters of mercury (mmHg). Reflects ocular and cerebrovascular dynamics.
Differences between groups in retinal vascular density (OCTA) | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Retinal vascular density measured using Optical Coherence Tomography Angiography (OCTA). Reported as percentage of perfused area in superficial and deep retinal layers.
Differences between groups in Peak systolic velocity of the ophthalmic artery | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Peak systolic velocity (PSV) of the ophthalmic artery will be measured by Doppler ultrasound. Values are expressed in centimeters per second (cm/s). Higher values may reflect increased arterial flow.
Differences between groups in End-diastolic velocity of the ophthalmic artery | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  End-diastolic velocity (EDV) of the ophthalmic artery will be measured by Doppler ultrasound. Values are expressed in centimeters per second (cm/s).
Differences between groups in Resistive index of the ophthalmic artery | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  The resistive index (RI) of the ophthalmic artery will be calculated using Doppler ultrasound as (PSV - EDV) / PSV. The RI is a dimensionless value ranging from 0 to 1, with higher values typically indicating increased vascular resistance.
Differences between groups in gut microbiota and intestinal permeability biomarkers | Baseline and 6-month follow-up.
  Gut microbiota is assessed using 16S rRNA sequencing. Permeability markers include zonulin (ZO-1) and lipopolysaccharide-binding protein (LBP).
Differences between groups in lipid profile | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Serum levels of total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglycerides will be measured. Values will be reported in mg/dL. Lower LDL and triglycerides, and higher HDL, are considered more favourable cardiovascular risk profiles.
Differences between groups in apolipoproteins and lipoprotein(a) | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Apolipoprotein B (ApoB), apolipoprotein A1 (ApoA1), and lipoprotein(a) [Lp(a)] will be measured. Units will be reported as mg/dL or nmol/L, depending on the marker. Higher ApoB and Lp(a) levels indicate greater cardiovascular risk, while higher ApoA1 is considered protective.
Differences between groups in liver function enzymes | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Plasma activities of alanine aminotransferase (ALT), aspartate aminotransferase (AST) and γ-glutamyl transferase (GGT) will be measured by standard kinetic assays. Results are expressed in U/L; lower values indicate better liver function.
Differences between groups in fasting insulin levels | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Serum insulin concentration will be determined by chemiluminescent immunoassay and reported in µU/mL; lower values reflect better insulin sensitivity.
Differences between groups in fasting glucose | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Plasma glucose will be measured by the hexokinase method and expressed in mg/dL.
Differences between groups in glycated haemoglobin | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Glycated haemoglobin will be analysed and reported as percentage of total haemoglobin (%); lower percentages indicate better long-term glycaemic control. Only for prediabetic and diabetic participants.
Differences between groups in renal function markers | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Serum urea, creatinine and uric acid will be measured by enzymatic assays and reported in mg/dL.
Differences between groups in glomerular filtration rate (GFR) | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  GFR will be calculated and expressed in mL/min/1.73 m²; higher values denote better kidney function.
Differences between groups in albuminuria | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Urinary albumin-to-creatinine ratio will be determined and reported in mg/g creatinine; lower values indicate better renal integrity.
Differences between groups in serum electrolytes | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Serum sodium, potassium and calcium will be quantified and expressed in mmol/L.
Differences between groups in leptin levels | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Serum leptin will be measured and reported in ng/mL.
Differences between groups in cortisol levels | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Serum cortisol will be determined and expressed in µg/dL.
Differences between groups in thyroid-stimulating hormone (TSH) | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Serum TSH will be analysed by immunoassay and reported in mIU/L.
Differences between groups in creatine phosphokinase (CPK) | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Serum CPK will be measured and expressed in U/L.
Differences between groups in beta-hydroxybutyrate (BHB) | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Serum BHB will be quantified and reported in mmol/L.
Differences between groups in inflammatory cytokines | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Plasma levels of IL-1β, IL-6, TNF-α and IL-10 will be determined using commercial ELISA kits. Values are expressed in pg/mL; lower pro-inflammatory (IL-1β, IL-6, TNF-α) and higher anti-inflammatory (IL-10) levels are considered favourable.
Differences between groups in brain-derived neurotrophic factor (BDNF) | Baseline, post-intervention (12 weeks), and 6-month follow-up.
  Serum BDNF will be quantified and reported in ng/mL; higher concentrations may reflect enhanced neuroplasticity.

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Spain

IPD SHARING:
Plan to Share IPD: No